CLINICAL TRIAL: NCT05444647
Title: Gut Microbiome Components Predict Response to Neoadjuvant Therapy in HER2-positive Breast Cancer Patients : A Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20210601
Record Dates: First submitted 2022-06-23; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: HER2-positive; neoadjuvant; microbiome
MeSH Terms: conditions — Breast Neoplasms | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — stool and blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HER2-positive: patients with newly diagnosed early stage HER2-positive breast cancer with an indication for standard trastuzumab-containing neoadjuvant treatment.
  Interventions: Procedure: stool and blood collection

INTERVENTIONS:
Procedure: stool and blood collection — Patients will collect fecal and blood samples prior to treatment and at the time of response evaluation, and completion of therapy using a standard stool-collection-kit. At the day of stool sampling, patients fill out a brief questionnaire about established factors that can change the microbiome such concurrent use of antibiotics and proton pump inhibitors.

SUMMARY:
In this study the characteristics and alterations of the gut microbiome during neoadjuvant therapy for HER2-positive breast cancer patients are studied, as well as the relation between the gut microbiome and probability of pCR.

DETAILED DESCRIPTION:
Although systemic treatment for early stage HER2-positive breast cancer is becoming increasingly effective, resistance and side effects of current treatment modalities are substantial. There is an urgent need for novel therapies, and in addition, better predictive tools are needed to select the right drug to the right patient. New data suggest that modulation of the microbiome of the gut might provide opportunities to increase anti-tumor efficacy of cancer therapies.

A better understanding of the composition, function and dynamics of the gut microbiome before and during trastuzumab-containing neoadjuvant treatment might help to identify factors that can be influenced during the treatment of patients with primary HER2-positive BC .

This study will prospectively enroll 100 participants with newly diagnosed HER2-positive breast cancer patients undergoing standard of care trastuzumab-containing neoadjuvant treatment and correlate gut microbiome composition with pCR.

Patients will be treated with the standard of care neoadjuvant therapy. Stool and peripheral blood (PB) samples will be collected at time of consent for therapy, mid-treatment, after the completion of neoadjuvant treatment (at the discretion of the medical oncologist). Correlation of changes in gut microbiome and metabolic changes, as well as inflammation and microbiome metabolites, will be assessed and possible connection with pCR and side effects will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Female, presenting for the first time with operable breast cancer, who had not received any previous treatment for an invasive malignancy.
2. Primary tumor greater than (>) 2 cm in diameter.
3. Age ≥ 18 years and < 70 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (</=) 1.
5. Baseline left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 55%
6. Availability of tumor tissue specimen after surgery.
7. Histologically proven diagnosis of breast cancer.
8. Patients have HER2-positive disease. HER2-positive disease was defined as follows: disease which overexpresses HER-2 by immunohistochemistry (IHC) 3+ and/or has HER2 amplification according to fluorescence in situ hybridization (FISH).
9. Had hormonal receptors (ER and PgR) assessed.
10. Signed informed consent.
11. Able to comply with the protocol.

Exclusion Criteria:

1. prior ipsilateral breast surgery, ipsilateral radiotherapy, hormonal therapy or systemic chemotherapy
2. Prolonged antibiotic treatment > 10 days within 1 month of neoadjuvant chemotherapy as prevention or suppression of an ongoing infection
3. Uncontrolled inflammatory bowel disease
4. pregnant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: early stage HER2-positive breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response in the breast and lymph nodes (ypT0/Tis ypN0) | 2 years
  The primary objective of this study is to determine if the probability of pCR (pathologic complete response) in HER2-positive breast cancer patients treated with standard of care neoadjuvant therapy is correlated with variability in the composition of intestinal microbiota and subsequent short-term alterations in that composition.

SECONDARY OUTCOMES:
Correlations between Pathologic complete Response | 2 years
  Determine if specific microbiota correlated with the probability of pCR are associated with the anti-tumor innate and adaptive immune responses in the peripheral blood
Side effects | 2 years
  Correlation of the microbiome to incidence of at least grade 3 toxicity using the CTCAE version 4.0 scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China